CLINICAL TRIAL: NCT00133497
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase II Study to Assess the Safety and Efficacy of the Cytomegalovirus gB/MF59 Vaccine in Preventing Systemic Cytomegalovirus Infection in Healthy Adolescent Females
Brief Title: gB/MF59 Vaccine in Preventing Cytomegalovirus Infection in Healthy Adolescent Females
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-039
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2013-09

CONDITIONS: Cytomegalovirus Infections
Keywords: cytomegalovirus, vaccine, women, children, parent protocol
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 20 mcg CMV gB + MF59 (Experimental): 200 subjects will receive vaccine CMV gB + MF59.
  Interventions: Biological: MF-59; Biological: CMV gB vaccine
- Saline (Placebo Comparator): 200 subjects will receive saline placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: MF-59 — Microfluoridized adjuvant 59 (MF59).
  Arms: 20 mcg CMV gB + MF59
Drug: Placebo — 0.5 mL of saline placebo.
  Arms: Saline
Biological: CMV gB vaccine — CMV glycoprotein B (gB) delivered as 20 mcg in 0.5 mL of vaccine.
  Arms: 20 mcg CMV gB + MF59

SUMMARY:
The purpose of this research study is to test the safety of and the body's response to an experimental cytomegalovirus (CMV) vaccine (called gB/MF59 vaccine). Participants will include approximately 400 healthy females, ages 12-17, recruited from adolescent clinics at Cincinnati Children's Hospital Medical Center, Vanderbilt University Medical Center, Baylor College of Medicine, University of Texas School of Public Health, Houston, and the University of Texas Medical Branch at Galveston. Participants will receive 3 doses of vaccine or placebo (saltwater) on a 0, 1, and 6 month schedule. Study procedures will include blood and urine samples. Participants will complete a diary recording temperatures and any side effects experienced. Subjects will be involved in study related procedures for up to 31 months.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, phase II study to assess the safety and efficacy of the cytomegalovirus glycoprotein B (gB)/MF59 vaccine in preventing systemic cytomegalovirus infection (CMV) in healthy adolescent females. The study interventions include: intramuscular (IM) injection of the investigational vaccine, CMV gB)/microfluidized adjuvant 59 (MF59), delivered as 20 micrograms in 0.5 mL of vaccine or IM injection of 0.5 mL of saline placebo. Subjects will be randomized (1:1) to receive vaccine or saline placebo. The primary efficacy objective is to assess whether injection with 3 doses of the CMV gB/MF59 vaccine will reduce the acquisition of a systemic CMV infection in healthy CMV-seronegative adolescent females. This will be accomplished by comparing the rates of acquisition of systemic CMV infection, defined as detection of CMV in the urine or blood, between the placebo and CMV vaccine recipients beginning 1 month after the third dose of vaccine. The primary safety objective is to assess the local and systemic effects of immunization and adverse events (AE) with the CMV gB/MF59 vaccine when administered to female adolescents on a 0-, 1-, and 6-month schedule. This will be assessed by comparing the rates of specific local and systemic reactogenicity events and AEs between the vaccine and placebo groups. The endpoint for this trial will be a systemic infection, which will be defined as identification of CMV from the urine (chosen because it is the most common site for isolation of CMV) or blood (chosen because it is the most likely route by which CMV reaches the fetus). Approximately 2400 healthy females, age 12 to 17 years (at time of initial enrollment) will be recruited in order to obtain approximately 400 CMV-seronegative subjects for the vaccine trial. Collection of sera will occur at Screening, Study Day 0, Month 6, Month 7 and every 3 months after Month 7. Collection of urine will occur at Study Day 0, Month 1, Month 2, Month 6, Month 7 and every 3 months after Month 7. Safety/reactogenicity monitoring will consist of solicited signs and symptoms self-reported by memory aid on the day of vaccination and for 6 follow-up days. Unsolicited symptoms will be collected for the 30-day period (± 2 days) after each vaccination and followed to adequate resolution or stabilization. The study duration for each subject will be 31 months: 7 months on the study with 24 months of follow-up beginning 1 month after the last injection. There will be 14 scheduled visits. This study is linked to DMID protocol 06-0043.

ELIGIBILITY:
Inclusion Criteria:

Subject Inclusion Criteria (Screening):

* Subjects must be willing and able to provide written informed assent prior to study enrollment; parent(s) or legal guardian must provide written informed consent prior to study enrollment.
* Subjects must be female and be 12 to 17 years at time of screening.
* Subjects must be willing to consider participation in the experimental cytomegalovirus (CMV) vaccine portion of the study which is 31-months in duration and must not be planning to relocate from the study area.
* Subjects must be using or willing to consider using effective methods of birth control. This includes abstinence or if sexually active using an effective method of birth control (e.g., oral contraceptives; diaphragm or condom in combination with contraceptive jelly; cream or foam; intrauterine contraceptive device; Depo-Provera®; skin patch; vaginal ring or cervical cap) for 30 days prior to vaccination and must agree to continue such precautions for 3 months after completion of the vaccination series.
* Subjects who are of childbearing potential must be willing to have a urine or serum pregnancy test within 24 hours before vaccination. The results will need to be negative to enroll in the vaccine study.

Subject's inclusion criteria (vaccine):

* Subject is willing and able to provide written informed assent prior to study enrollment; parent(s) or legal guardian provides written informed consent prior to study enrollment.
* Subject is female and 12 to 17 years at time of screening.
* Subject is available for the 31-month duration of the study (7 months on the study and 24 months of follow-up beginning 1 month after the last injection) and is not planning to relocate from the study area.
* Subject must agree to practice abstinence, or if sexually active must be using an effective method of birth control (e.g., oral contraceptives; diaphragm or condom in combination with contraceptive jelly; cream or foam; intrauterine contraceptive device; Depo-Provera®; skin patch; vaginal ring or cervical cap) for 30 days prior to vaccination and must agree to continue such precautions for 3 months after completion of the vaccination series.
* Subject of child bearing potential has a negative urine or serum pregnancy test within 24 hours of vaccination.
* Subject is willing and able to comply with the requirements of the protocol (e.g., completion of the memory aid, return for follow-up visits, accessible by phone and not planning on moving from the study area).

Subject Inclusion Criteria (Shedding):

* Subjects must be willing and able to provide written informed assent prior to study enrollment; parent(s) or legal guardian must provide written informed consent prior to study enrollment.
* Subject is positive for antibodies to CMV detected by enzyme-linked immunosorbent assay (ELISA) using a commercial CMV antibody assay screen.
* Subjects must be willing and able to comply with the requirements of the protocol (e.g., completion of the visits, accessible by phone and not planning on moving from the study area).

Exclusion Criteria:

Subject Exclusion Criteria (Screening):

* Receipt of blood and/or blood products in the past 3 months
* Known to be pregnant or lactating
* Planning to become pregnant during the first 8 months of the study (Months 0-8);
* Known previous infection with cytomegalovirus (CMV);
* Previously received a CMV vaccine;
* History of allergic reactions to any component of the study vaccine;
* History of malignancy or have a confirmed or suspected immunodeficient condition, such as human immunodeficiency virus (HIV) infection;
* History of current acute or chronic autoimmune disease;
* History of ongoing clinically significant illness (diabetes, pulmonary, cardiovascular, hepatic or renal functional abnormality) as determined by medical history;
* History of any neurologic disorders or seizures, with the exception of febrile seizures during childhood;
* Presently receiving or history of receiving any medications or treatments that affect the immune system such as immune globulin, interferon, immunomodulators, cytotoxic drugs or drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable) in the past 6 months. Inhaled and topical corticosteroids will be allowed;
* History of depression not controlled with current drug therapy or involving institutionalization;
* History of schizophrenia or psychosis;
* History of suicide attempt;
* Active substance or alcohol abuse;
* Currently enrolled in another research study. (Subjects participating in a non-interventional studies, questionnaires, or observational studies will not be excluded from participation).

Subjects exclusion criteria (vaccine):

* Antibodies to CMV that are detected at the screening visit;
* Previously received a CMV vaccine;
* Subject is planning on becoming pregnant during the first 8 months of the vaccine study;
* Subject receives an experimental drug or vaccine in the 30 days prior to the first dose of vaccine or planned receipt before 30 days after the final dose of the vaccine;
* Subject receives or is planning to receive a nonstudy vaccine within 30 days before or after any dose of study vaccine with the following exceptions: Administration of routine meningococcal, hepatitis A, hepatitis B, Tdap (Tetanus, Diphtheria, Pertussis), human papillomavirus (HPV), inactivated influenza (but not FluMist®), diphtheria/tetanus and/or diphtheria/tetanus-containing vaccine up to 8 days before or at least 8 days after a dose of study vaccine is allowed. Administration of vaccine injection can be delayed if a nonstudy vaccine has been administered and will be given as soon as acceptable;
* Subject has an acute disease within 72 hours prior to enrollment in the vaccine study, defined as the presence of a moderate or severe illness (as determined by the investigator through medical history and physical examination. Study vaccine can be administered to persons with a minor illness, such as diarrhea, or mild upper respiratory tract infection with or without low-grade febrile illness. Vaccination can be delayed until the subject has recovered;
* Subject receives systemic corticosteroids > 2mg/kg for >14 days. Inhaled and topical steroids are permitted.

Subject Exclusion Criteria (Shedding):

None

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 409 (Actual)
Dates: Start 2006-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Efficacy: systemic cytomegalovirus (CMV) infection, defined by the detection of CMV in the urine or blood, which will be evaluated by CMV detection by polymerase chain reaction (PCR). | Study Day 0, Month 1, Month 2, Month 6, Month 7 and every 3 months after Month 7.
Safety: incidence of local and systemic reactions, as determined by self-reported assessments using a memory aid, adverse events (AEs) and serious adverse events (SAEs). | Local and systemic reactions within 7 days of vaccination; adverse events (AEs) within the 30 day period after vaccination; serious adverse events (SAEs) observed any time throughout the duration of study.

SECONDARY OUTCOMES:
Efficacy: CMV infections defined as seroconversion to nonvaccine CMV antigens or identification of CMV in the blood or urine. | Specimens collected every 3 months.
Immunologic: CMV antibody measurements by CMV neutralization, enzyme-linked immunosorbent assay (ELISA), and CMV glycoprotein B (gB) assay. | Study Day 0, Month 6, Month 7 and every 3 months after Month 7.
Duration and magnitude of CMV replication in the urine and blood as determined from specimens. | Obtained monthly for 4 months and then every other month for 8 months after identification of CMV infection.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee
  - The University of Texas Medical Branch - Sealy Center for Vaccine Development (SCVD), Galveston, Texas
  - The University of Texas Health Science Center - Pediatrics, Houston, Texas
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas

REFERENCES:
- [Derived] Hu X, Karthigeyan KP, Herbek S, Valencia SM, Jenks JA, Webster H, Miller IG, Connors M, Pollara J, Andy C, Gerber LM, Walter EB, Edwards KM, Bernstein DI, Hou J, Koch M, Panther L, Carfi A, Wu K, Permar SR. Human Cytomegalovirus mRNA-1647 Vaccine Candidate Elicits Potent and Broad Neutralization and Higher Antibody-Dependent Cellular Cytotoxicity Responses Than the gB/MF59 Vaccine. J Infect Dis. 2024 Aug 16;230(2):455-466. doi: 10.1093/infdis/jiad593. PMID 38324766